CLINICAL TRIAL: NCT06320132
Title: BLANDISH (Brain, Loss of Function, Aneurism, Disease, Injury, Stroke, Hemorrhage): Design and Internal Validation of an AI System to Support and Optimize the Management of Spontaneous Intracranial Hemorrhage Patients in the NeuroICU
Brief Title: BLANDISH (Brain, Loss of Function, Aneurism, Disease, Injury, Stroke, Hemorrhage)
Acronym: BLANDISH
Status: Recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Francesca Guzzo, Principal Investigator, IRCCS Ospedale San Raffaele
Other Study IDs: BLANDISH
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Intracranial Hemorrhages
MeSH Terms: conditions — Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 14 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective group: Patients treated for spontaneous intracranial hemorrhage before March 13, 2024.
  Interventions: Other: Treatment of spontaneous intracranial hemorrhage
- Prospective group: Patients treated for spontaneous intracranial hemorrhage after March 13, 2024.
  Interventions: Other: Treatment of spontaneous intracranial hemorrhage

INTERVENTIONS:
Other: Treatment of spontaneous intracranial hemorrhage — Data collection of therapeutic approach, including radiological, medical, surgical therapies.

SUMMARY:
The goal of this observational study is to train a machine learning system based on data from patients affected by spontaneous Intracranial Hemorrage. The main question it aims to answer is whether there is a correlation between actual clinical pratice, reached outcomes and favorable or unfavorable predictive factors, and anamnesis.

Participants will be treated as per standard clinical practice.

DETAILED DESCRIPTION:
In NeuroICU, treatments typically adhere to guidelines based on scientific consensus. Despite this, the prognosis for patients with intracranial hemorrhages has not significantly improved over recent decades, resulting in generally unsatisfactory outcomes. While randomized controlled trials (RCTs) are considered the gold standard for clinical research, they can be expensive and ethically challenging to conduct. Observational studies provide an alternative method, offering larger datasets covering longer periods, which can be more beneficial and feasible for certain research endeavors.

Machine Learning (ML) algorithms, unlike classical statistical methods, have the capability to process a vast number of variables, offering a personalized and dependable approach for healthcare providers in patient management. Recognizing the necessity for well-designed studies to identify optimal therapeutic strategies for neurocritical patients and acknowledging the limitations of existing guidelines, we aim to leverage ML programs to develop an advanced system capable of uncovering data patterns and linking them to potential outcomes.

The BLANDISH project focuses on patients with spontaneous intracerebral hemorrhage (sICH), a condition lacking proven beneficial treatment. By collecting and analyzing data from sICH patients admitted to neuroICU, the project aims to develop a supervised ML algorithm named BLANDISH.

This algorithm will stratify patients based on prognosis, identifying those at highest risk of death and secondary brain injuries. By guiding each patient towards the most targeted therapeutic strategy, the algorithm could help improve patient outcomes and assess the effectiveness of current clinical practices. Additionally, it may enable healthcare staff to better allocate resources and introduce individualized therapeutic programs based on precision medicine, potentially reducing hospitalization times and healthcare costs.

The initial step in developing the BLANDISH algorithm involves collecting clinical data, stored in a structured datalake, which serves as a data repository. This platform will gather information on the clinical course of sICH patients admitted to neuroICU. After data collection, the next steps include preprocessing, variable selection correlated with patient mortality, and algorithm training with input data and internal validation to control its behavior. External validation will follow, involving data collection from various clinical centers to assess the algorithm's reliability and generalization capacity. A multicenter observational clinical study will then be conducted to validate the BLANDISH algorithm, aiming to determine its impact on sICH patient outcomes. This final phase includes a survival study comparing patients in the experimental group (whose treatment is guided by BLANDISH) with those following standard clinical practice. The project aims to demonstrate the superiority of the ML approach over current guidelines, evaluating the accuracy and potential improvements in patient management across different care settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients who enter the NICU for acute spontaneous intracranial hemorrhage
* Adult patients (≥ 18 years)
* Sex: female, male, intersex

Exclusion Criteria:

* All patients affected by non-spontaneous ICH
* Patients with sICH determined by brain tumor or brain metastases
* All patients affected by chronic ICH
* Pregnant and puerperal women
* Refusal to participate in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients affected by spontaneous Intracranial Hemorrhage.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 12 months
  Patients who die within 12 months after being treated for spontaneous intracranial hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Guzzo, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No